CLINICAL TRIAL: NCT02951338
Title: Promoting Optimal Physical Exercise for Life (PROPEL) - Aerobic Exercise and Self-management Early After Stroke to Increase Daily Physical Activity: a Randomized Trial
Brief Title: PROPEL Randomized Trial
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 pandemic
Sponsor: Toronto Rehabilitation Institute (Other)
Collaborators: Sunnybrook Research Institute (Other); West Park Healthcare Centre (Other); Hamilton Health Sciences Corporation (Other); McMaster University (Other); St. Joseph's Care Group (Other)
Responsible Party: Principal Investigator, Avril Mansfield, Principal Investigator, Toronto Rehabilitation Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 16-5916
Record Dates: First submitted 2016-10-25; First posted 2016-11-01 (Estimated); Results first posted 2025-04-11 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Stroke
Keywords: Physical activity; Exercise; Behaviour change; Rehabilitation; Self-management; Education
MeSH Terms: conditions — Stroke; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group aerobic exercise only (Active Comparator): Supervised group exercise up to 3-times/week for 6 weeks. A typical exercise session will involve a 3-5 minute 'warm-up', 20-30 minutes of aerobic exercise at a target heart rate determined from a sub-maximal test, and a 3-5 minute 'cool-down' of low-intensity exercise. The choice of exercise modality for the submaximal test and for training (e.g., recumbent stepper, cycle ergometer, or treadmill) will be individually prescribed based on patients' sensori-motor recovery, postural control, functional abilities, and safety. Heart rate, blood pressure, rate of perceived exertion, workload, and duration of training will be documented for each session. These data will be reviewed by the physiotherapist with appropriate progression of the intensity and/or duration of exercise as necessary.
  Participants may receive general advice to keep physically active after discharge, and may receive an individualized home exercise program, as is currently routine care at all sites.
  Interventions: Other: Group aerobic exercise
- PROPEL program (Experimental): The PROPEL program involves both group aerobic exercise (as described above) and group discussion aimed at enabling participation in exercise after discharge. Components of the PROPEL program were developed according to the Transtheoretical Model of health behaviour change and Social Cognitive Theory. In addition to group exercise participants will attend 1-hour small group discussion sessions once weekly to learn self-management skills for exercise in preparation for discharge from rehabilitation. These discussions include: identifying and solving problems around barriers to exercise; understanding personal and general benefits of exercise; exploring appropriate community resources for exercise; and finding individualized and realistic strategies for incorporating exercise in a regular routine. Participants will become comfortable with progressing their exercise and will set short- and long-term exercise goals.
  Interventions: Behavioral: PROPEL program

INTERVENTIONS:
Behavioral: PROPEL program — The PROPEL program involves both group aerobic exercise and group discussion aimed at enabling participation in exercise after discharge. Components of the PROPEL program were developed according to the Transtheoretical Model of health behaviour change and Social Cognitive Theory. In addition to group exercise participants will attend 1-hour small group discussion sessions once weekly to learn self-management skills for exercise in preparation for discharge from rehabilitation. These discussions include: identifying and solving problems around barriers to exercise; understanding personal and general benefits of exercise; exploring appropriate community resources for exercise; and finding individualized and realistic strategies for incorporating exercise in a regular routine. Participants will become comfortable with progressing their exercise and will set short- and long-term exercise goals.
  Arms: PROPEL program
Other: Group aerobic exercise — Supervised group exercise up to 3-times/week for 6 weeks. A typical exercise session will involve a 3-5 minute 'warm-up', 20-30 minutes of aerobic exercise at a target heart rate determined from a sub-maximal test, and a 3-5 minute 'cool-down' of low-intensity exercise. The choice of exercise modality for the submaximal test and for training (e.g., recumbent stepper, cycle ergometer, or treadmill) will be individually prescribed based on patients' sensori-motor recovery, postural control, functional abilities, and safety. Heart rate, blood pressure, rate of perceived exertion, workload, and duration of training will be documented for each session. These data will be reviewed by the physiotherapist with appropriate progression of the intensity and/or duration of exercise as necessary.
  Participants may receive general advice to keep physically active after discharge, and may receive an individualized home exercise program, as is currently routine care at all sites.
  Arms: Group aerobic exercise only

SUMMARY:
It is important for people with stroke to exercise in order to improve their overall recovery and general health. However, these individuals are less physically active than people without stroke, and they often do not achieve the recommended frequency, intensity or duration of exercise. Low levels of physical activity leads to people with stroke becoming very unfit, which can result in functional decline and increased difficulty being active. It is important to determine how to encourage people with stroke to be more active in the long-term. The transition time between the end of rehabilitation and return to the community might be an ideal time to address barriers, and to develop positive habits, knowledge and abilities for long-term participation in exercise. We developed the PROPEL program that combines exercise with self-management strategies during rehabilitation to promote physical activity after rehabilitation. Preliminary pilot findings indicate that people who completed PROPEL were more physically active after discharge than those who did not. This study aims to evaluate the effect of PROPEL on long-term participation in exercise after discharge from stroke rehabilitation. This study will take place at 6 different hospitals. Participants will either complete a control intervention (group exercise only) or the PROPEL intervention (group exercise plus self-management). Participants' adherence to exercise for 6 months after the end of the interventions will be evaluated using activity and heart rate monitors and physical activity questionnaires. We expect this study will show that a simple intervention delivered during rehabilitation will increase participation in exercise after rehabilitation. Increased participation in exercise could then lead to improved stroke recovery and overall health, and reduced risk of having another stroke.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who are referred to the group aerobic exercise or PROPEL programs as part of their stroke rehabilitation.

Exclusion Criteria:

* Language or communication barrier that prevents completion of questionnaires (e.g., severe receptive or global aphasia or non-English speaking);
* Cognitive impairment that would prevent participation in unsupervised exercise;
* Attend less than 50% of group aerobic exercise/PROPEL sessions; and/or
* Attend less than 4 of the 6 group discussion sessions (for individuals referred to the PROPEL program).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2020-09-13 (Actual); Study Completion 2020-09-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Avril Mansfield, PhD, Principal Investigator — Toronto Rehabilitation Institute - UHN
Locations (5):
- Canada (5):
  - Hamilton Health Sciences, Hamilton, Ontario
  - St. Joseph's Care Group, Thunder Bay, Ontario
  - Sunnybrook Research Institute, Toronto, Ontario
  - West Park Healthcare Centre, Toronto, Ontario
  - Toronto Rehabilitation Institute - UHN, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mansfield A, Knorr S, Poon V, Inness EL, Middleton L, Biasin L, Brunton K, Howe JA, Brooks D. Promoting Optimal Physical Exercise for Life: An Exercise and Self-Management Program to Encourage Participation in Physical Activity after Discharge from Stroke Rehabilitation-A Feasibility Study. Stroke Res Treat. 2016;2016:9476541. doi: 10.1155/2016/9476541. Epub 2016 May 30. PMID 27313948
- [Result] Devasahayam AJ, Tang A, Taylor D, Inness EL, Fleck R, French E, Jagroop D, Danells CJ, Mansfield A. Cardiorespiratory exercise and self-management early after stroke to increase daily physical activity: results from a stepped-wedge cluster randomised trial. Disabil Rehabil. 2025 Jul;47(14):3581-3591. doi: 10.1080/09638288.2024.2426689. Epub 2024 Nov 12. PMID 39530472
- [Derived] Mansfield A, Brooks D, Tang A, Taylor D, Inness EL, Kiss A, Middleton L, Biasin L, Fleck R, French E, LeBlanc K, Aqui A, Danells C. Promoting Optimal Physical Exercise for Life (PROPEL): aerobic exercise and self-management early after stroke to increase daily physical activity-study protocol for a stepped-wedge randomised trial. BMJ Open. 2017 Jun 30;7(6):e015843. doi: 10.1136/bmjopen-2017-015843. PMID 28667222

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group Aerobic Exercise Only | PROPEL Program
Started | 28 | 29
1-month Follow-up | 26 | 23
4-month Follow-up | 24 | 16
Completed | 22 | 16
Not Completed | 6 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group Aerobic Exercise Only | PROPEL Program | Total
Number analyzed (Participants) | 28 | 29 | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.9 (13.6) | 61.7 (13.5) | 60.8 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 12 | 26
  Male | 14 | 17 | 31
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Time post-stroke [Mean (Standard Deviation); unit: days] — Time post-stroke at study enrollment
  days | 129 (83) | 106 (66) | 117.8 (74.9)
More affected side [Count of Participants; unit: Participants]
  Left | 15 | 13 | 28
  Right | 11 | 13 | 24
  Both | 1 | 3 | 4
  Neither | 1 | 0 | 1
Type of stroke [Count of Participants; unit: Participants]
  Infarct | 19 | 22 | 41
  Hemorrhage | 8 | 6 | 14
  Unknown | 0 | 1 | 1
  Other | 1 | 0 | 1
Chedoke-McMaster Stroke Assessment [Mean (Standard Deviation); unit: score] — Motor impairment scale. Scale range: 1-7. Lower values indicate greater motor impairment.
  score
    Leg | 5.2 (1.2) | 5.0 (4.8) | 5.1 (1.2)
    Foot | 5.0 (1.8) | 4.8 (1.2) | 4.9 (1.6)
National Institutes of Health Stroke Scale [Mean (Standard Deviation); unit: score] — Measure of stroke severity. Scale range: 0-42. Higher values indicate more severe strokes.
  score | 3.4 (3) | 3.3 (2.7) | 3.3 (2.8)
Montreal Cognitive Assessment [Mean (Standard Deviation); unit: score] — Cognitive function assessment. Scale range: 0-30. Higher values indicate greater cognitive function.
  score | 23.3 (4.9) | 24.1 (4.5) | 23.7 (4.7)
Pre-morbid moderate or strenuous occupation [Count of Participants; unit: Participants] | 17 | 18 | 35
Pre-morbid time in active transportation [Mean (Standard Deviation); unit: hours/week] | 6.3 (8.6) | 7.6 (10.4) | 7.0 (9.5)
Pre-morbid exercise participation [Count of Participants; unit: Participants] | 20 | 18 | 38
Pre-morbid time spent exercising [Mean (Standard Deviation); unit: hours/week] | 1.8 (2.6) | 1.8 (4.0) | 1.8 (3.4)

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Meet Recommended Intensity, Frequency, and Duration of Physical Activity
Description: The primary outcome is proportion of participants per group who meet recommendations for intensity, frequency, and duration of daily physical activity; that is, at least 150 minutes per week of moderate-to-vigorous intensity exercise. Physical activity will be assessed using a step counter, heart rate monitor, and questionnaire for 7 continuous days.
  Participants will be deemed to meet the recommendations within a given week if they meet at least two of three criteria at 6-months post-discharge: 1) record at least 150 'active minutes' (from the step activity monitor); 2) record at least 150 minutes of heart rate between 55-80% of age-predicted maximum; and/or 3) report at least 150 minutes of moderate and/or vigorous intensity activity on the physical activity questionnaire.
Time Frame: 6-months post-discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Group Aerobic Exercise Only | PROPEL Program
Number analyzed (Participants) | 22 | 17
Participants | 9 | 6

2. Secondary Outcome: Short Self-Efficacy for Exercise Scale
Description: 4-item self-efficacy for exercise scale. Scale range: 1-5. The total score is the mean of the scores of the individual items. Higher values represent better outcome.
Time Frame: 0-1 week post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group Aerobic Exercise Only | PROPEL Program
Number analyzed (Participants) | 28 | 28
score on a scale | 3.2 (0.8) | 3.8 (0.7)

3. Secondary Outcome: Short Outcome Expectation for Exercise Scale
Description: 5-item scale. Scale range: 1-5. The total score is the mean of the scores for the individual items. Higher values represent better outcome.
Time Frame: 0-1 week post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group Aerobic Exercise Only | PROPEL Program
Number analyzed (Participants) | 28 | 28
score on a scale | 4.3 (0.6) | 4.4 (0.5)

4. Secondary Outcome: Barriers to Being Active Quiz - Category Scores
Description: Scale range for each category: 0-12. Higher scores indicate greater reported barriers for that category. The category score is the sum of the individual item scores within each category.
Time Frame: 1 month post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group Aerobic Exercise Only | PROPEL Program
Number analyzed (Participants) | 22 | 21
score on a scale
  Time | 1.5 (1.5) | 2.1 (2.3)
  Influence | 1.6 (1.3) | 2.1 (1.8)
  Energy | 1.9 (2.0) | 2.0 (2.2)
  Willpower | 3.0 (2.5) | 2.0 (2.2)
  Injury | 1.4 (1.5) | 1.5 (2.2)
  Skill | 1.5 (1.9) | 1.5 (1.9)
  Facilities | 2.5 (2.5) | 1.8 (2.0)

5. Secondary Outcome: Barriers to Being Active Quiz - Number of Significant Barriers
Description: Scale range for number of significant barriers: 0-7. Number of significant barriers is the number of BBAQ categories with a score of 5 or higher. A higher value indicates worse outcome.
Time Frame: 1 month post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group Aerobic Exercise Only | PROPEL Program
Number analyzed (Participants) | 22 | 21
score on a scale | 0.9 (1.1) | 0.9 (1.4)

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Group Aerobic Exercise Only | PROPEL Program
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/29
Other Adverse Events (participants affected / at risk) | 0/28 | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-16): https://cdn.clinicaltrials.gov/large-docs/38/NCT02951338/Prot_SAP_000.pdf